CLINICAL TRIAL: NCT06231849
Title: Gut Microbiota Dysbiosis in Opioid Use Disorders: Implications for Clinical Symptoms and Relapse Rate.
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, ahmed mohammed abdelrahim, Resident doctor, Assiut University
Other Study IDs: gut microbiota in opioid use
Record Dates: First submitted 2023-12-27; First posted 2024-01-30 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Opioid Use; Opioid Use Disorder; Opioid Dependence
Keywords: gut microbiota .; Opioid use
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Occult Blood

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — stool analysis to determine the number of gut microbiota in individuals with opioid use disorders.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- normal subjects without opioid intoxications.: 1. Individuals of male gender aged between 20 to 35 years old
- individuals with opioid use disorders.: Individuals of male gender aged between 20 to 35 years old with opioid use disorders.
  Interventions: Diagnostic Test: stool analysis

INTERVENTIONS:
Diagnostic Test: stool analysis — stool analysis to determine number of gut microbiota in subjects with opioid use and its effect on its intoxication.
  Groups: individuals with opioid use disorders.

SUMMARY:
This study will aim to investigate the gut microbiota in Egyptian patients with opioid use disorders and correlate microbiota bacterial abundance with clinical data.

DETAILED DESCRIPTION:
Addiction is defined as a chronic, relapsing disorder characterized by compulsive drug seeking and use despite adverse consequences. Pathological substance use disorders represent a major public health crisis with limited effective treatment options. Although the gut and brain are separate organs, they communicate with each other via trillions of intestinal bacteria that collectively make up one's gut microbiome. Findings from both humans and animals support a critical role of gut microbes in regulating brain function, mood, and behavior. Gut bacteria influence neural circuits that are notably affected in addiction-related behaviors. These include circuits involved in stress, reward, and motivation, with substance use influencing gut microbial abnormalities, suggesting significant gut-brain interactions in drug addiction.

The investigator will discuss this role of gut microbiome in Assuit university hospital to see how the pathogenesis can be altered of drug addiction.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical and laboratory diagnosis of substance missuse.
2. Must be encountering withdrawal symptoms for the first time.

Exclusion Criteria:

1. An intelligence quotient (IQ) below 70.
2. Gastrointestinal diseases.

Ages: 20 Years to 35 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — biological sex
Study Population: Patients in the intoxication stage of addiction will be initially included and undergo a comprehensive psychiatric and medical assessment. This assessment will be repeated one month later when patients transition into the withdrawal stage, and finally, a follow-up assessment will occur three months later. On the other hand, healthy control group will be matched in age and gender will be recruited.
Sampling Method: Probability Sample
Enrollment: 52 (Estimated)
Dates: Start 2024-02 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Determine the psychiatric symptoms related to opioid misuse. | 3 months.
  The investigator will focus on the following scale:
  • The Symptom ChickList-90-Revised : psychiatric Symptom related to opioid misuse measured by symptom checklist.
Determine severity of misuse. | 3 months.
  Addiction severity index: is an assessment tool used to assess an adult's condition in 7 key problem areas that are typically affected by substance abuse, including medical status, employment, and more, it addresses 7 main aspects of a person's behavior and environment.1 The areas assessed include:1
  Medical status. Employment and support. Drug use. Alcohol use. Legal status. Family/social status. Psychiatric status. substance abuse assessment uses the composite score to assign a severity rating. The ratings are based on a scale of 0 to 9 as follows: 0-1: No imminent problem, treatment not indicated. 2-3: Slight problem; treatment may not be necessary. 4-5: Moderate problem, a treatment plan should be considered. 6-7: Considerable difficulty, begin a treatment plan. 8-9: Extreme problem, treatment is vital.
Determine type of misuse(whether its just opioid or combined with other substances) | 3 months
  • Laboratory: Urine analysis for substance use(drug screen).

SECONDARY OUTCOMES:
Measuring abundance of gut microbiota | 6 months
  The investigator will perform a stool analysis to determine changes in amount of gut microbiota in both intoxication phase and in recovery phase then after 3 month a follow-up test will be conducted to determine the percent of Relapse rate.

CONTACTS AND LOCATIONS:
Overall Officials: Alaa El-Din Darwish Othman, professor, Study Chair — assiutbird25@aun.edu.eg; GeLLan Karamallah Ramadan, doctor, Study Director — gillankaram@aun.edu.eg

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Acharya C, Betrapally NS, Gillevet PM, Sterling RK, Akbarali H, White MB, Ganapathy D, Fagan A, Sikaroodi M, Bajaj JS. Chronic opioid use is associated with altered gut microbiota and predicts readmissions in patients with cirrhosis. Aliment Pharmacol Ther. 2017 Jan;45(2):319-331. doi: 10.1111/apt.13858. Epub 2016 Nov 20. PMID 27868217
- [Background] Akbarali HI, Dewey WL. The gut-brain interaction in opioid tolerance. Curr Opin Pharmacol. 2017 Dec;37:126-130. doi: 10.1016/j.coph.2017.10.012. Epub 2017 Nov 13. PMID 29145012
- [Background] Berridge KC. From prediction error to incentive salience: mesolimbic computation of reward motivation. Eur J Neurosci. 2012 Apr;35(7):1124-43. doi: 10.1111/j.1460-9568.2012.07990.x. PMID 22487042